CLINICAL TRIAL: NCT05431309
Title: Role of Screening With Coronary Computed Tomography Angiography in Primary Prevention of Coronary Heart Disease: a Community-based, Prospective Randomised Controlled Study
Brief Title: Role of Screening With Coronary Computed Tomography Angiography in Primary Prevention of Coronary Heart Disease
Acronym: RESPECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhang longjiang,MD, Principal Investigator : Zhang longjiang, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZRui
Record Dates: First submitted 2022-06-03; First posted 2022-06-24 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Cardiovascular Primary Prevention Strategy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CCTA-based strategy group (Active Comparator): Patients will be managed following the CCTA -based coronary heart disease prevention strategy for statin initiation and follow-up.
  Interventions: Diagnostic Test: Coronary Computed Tomography Angiography
- Traditional strategy group (Sham Comparator): Patients will be managed following the Traditional cardiovascular disease prevention strategy based on Chinese guideline for statin initiation and follow-up.
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Diagnostic Test: Coronary Computed Tomography Angiography — Intervention strategies were selected according to CCTA results
  Arms: CCTA-based strategy group
Other: Standard Treatment — Traditional cardiovascular disease prevention strategy based on Chinese guideline
  Arms: Traditional strategy group

SUMMARY:
The primary objective of this study is to determine whether coronary computed tomography angiography (CCTA) -based coronary heart disease(CHD) prevention strategy will be superior to traditional CHD prevention strategy, in reducing the future risk of CHD which included myocardial infarction, angina, cardiac death, and an emergency/urgent coronary revascularisation procedure, in a community population aged 40 to 69 years with cardiovascular risk factors but no history of cardiovascular disease.

DETAILED DESCRIPTION:
Recent studies found that the incidence of CAD, screening with CCTA, in the general population is as high as 42%~49%. However, the effectiveness of CCTA screening in the primary prevention of CHD is unclear. The investigators designed a randomized controlled, open-label, pragmatic study to determine whether coronary computed tomography angiography (CCTA) -based coronary heart disease(CHD) prevention strategy will be superior to traditional CHD prevention strategy.

Community volunteers aged 40 to 69 years who provide consent, and are eligible (with cardiovascular risk factors but no history of cardiovascular disease), will be randomized 1:1 to receive individualized primary prevention programs for CHD, including statin recommendation, based on CCTA results or traditional risk assessment results using the Chinese guideline on the primary prevention of cardiovascular diseases-recommended strategy. All subjects will be followed for 5 years, but until the target primary endpoint event is met. The primary composite outcome was the first occurrence of CHD, which included myocardial infarction, angina, cardiac death, and an emergency/urgent coronary revascularisation procedure.

In order to prepare the study with high quality, the investigators will performed a pilot study prior to the initiation of patient recruitment for the main study.

ELIGIBILITY:
Inclusion Criteria:

1. Resident population aged 40-69 in Nanjing, China
2. One or more of the following cardiovascular disease risk factors must be present, as follows:

   1. Current or recent (within 12 months) smoker
   2. Clinical diagnosis of hypertension (>140/90mmHg)
   3. Hypercholesterolaemia (LDL≥4.1mmol/L or total cholesterol>6.0 mmol/L, including familial hypercholesterolaemia)
   4. Diabetes mellitus
   5. Rheumatoid arthritis
   6. Systemic lupus erythematosus
   7. Family history of premature cardiovascular disease (first degree relative with atherosclerotic cardiovascular disease, males, age<55 years; females, age<60 years)
   8. Chronic kidney disease stage 3 (eGFR 30~59mL/min/1.73 m2)

Exclusion Criteria:

1. Plan to leave Nanjing within 5 years or be unable to complete the follow-up work
2. Refuse to sign informed consent or inability to understand and comply with the program process
3. Known atherosclerotic cardiovascular disease (eg. angina, coronary heart disease, stroke, transient ischemic attack, peripheral vascular disease)
4. Serious chronic kidney disease (eGFR< 30 ml/min/1.73 m2)
5. Serious liver disease or dysfunction (chronic active hepatitis and cirrhosis, or aspartate aminotransferase (AST) or alanine transaminase (ALT) > 3 times the upper limit of normal)
6. Prior coronary computed tomography angiography or invasive coronary angiography within the last 5 years
7. Not appropriate to be tested due to birth planning, allergies, acute thyroid storm, etc
8. Current use of statin therapy
9. Patients with diseases that seriously affect the survival period, such as malignant tumors
10. Other conditions at the discretion of the research group

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15000 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
The first occurrence of coronary heart disease | 5 years
  Composite of cardiac death, myocardial infarction, angina, and an emergency/urgent coronary revascularisation procedure.

SECONDARY OUTCOMES:
Major cardiovascular adverse events (MACE) | 5 years
  Number of cardiac death, myocardial infarction, emergency/urgent coronary revascularisation procedure and stroke
Death | 5 years
  Number of all-cause death, cardiovascular deaths, non-cardiovascular deaths and undetermined death
Occurrence of serious adverse events related to iodinated contrast agent | 1 year
  Composite outcome: contrast-induced nephropathy and severe allergoid contrast agent reaction
Coronary interventions | 5 years
  Number of invasive coronary angiography and coronary revascularisation procedures
The primary end point(composite of cardiac death, myocardial infarction, angina, and an emergency/urgent coronary revascularisation procedure) in different subgroups | 5 years
  The primary end point(composite of cardiac death, myocardial infarction, angina, and an emergency/urgent coronary revascularisation procedure) will be analyzed in prespecified subgroups, including age, sex, diabetes, smoking status, hypertension, diabetes mellitus, hyperlipidemia, Chronic kidney disease stage 3
Diet | at 1-year follow-up and final follow-up (5 years)
  Measured by Food Frequency Questionnaire
Exercise | at 1-year follow-up and final follow-up (5 years)
  Change in activity levels measured through International Physical Activity Questionnaire(IPAQ)
Smoking cessation | at 1-year follow-up and final follow-up (5 years)
  Proportion of patients who changed smoking habits (%)
Change in cardiovascular risk factors (blood pressure) | at 1-year follow-up and final follow-up (5 years)
  Blood pressure(mmHg)
Change in cardiovascular risk factors (lipids) | at 1-year follow-up and final follow-up (5 years)
  Lipids(mmol/L)
Change in cardiovascular risk factors (body weight) | at 1-year follow-up and final follow-up (5 years)
  Body weight(kg)
Change in cardiovascular risk factors(waist circumference) | at 1-year follow-up and final follow-up (5 years)
  Waist circumference(cm)
Change in depression (PHQ-9) | at 1-year follow-up and final follow-up (5 years)
  Change in depression measured using Patient Health Questionnaire-9 (PHQ-9) instrument
Change in anxiety (GAD-7) | at 1-year follow-up and final follow-up (5 years)
  Change in anxiety measured using Generalized Anxiety Disorder 7-item (GAD-7) instrument
Change in quality of sleep(PSQI) | at 1-year follow-up and final follow-up (5 years)
  Change in quality of sleep measured using Pittsburgh Sleep Quality Index (PSQI) instrument
Change in quality of life(SF-12) | at 1-year follow-up and final follow-up (5 years)
  Change in quality of quality of life measured using 12-item Short-Form Health Survey Questionnaire (SF-12) instrument
Incidental findings in Computed Tomography Angiography group | at 1-year follow-up and final follow-up (5 years)
  Potential benefits and harms of the findings
Medication adherence( anti-hypertension agent, hypoglycemic agent, antilipemic agents, anti-platelet, etc.) | at 1-year follow-up and final follow-up (5 years)
  Measure adherence using follow-up questionnaires (Whether participants are taking medication, why participants are not taking it or taking it, the name, frequency, dosage and side effects of the medication participants are taking)
Health economics | 5 years
  Cost-Effectiveness analysis and Cost-Utility analysis
Disadvantages of Radiation exposure | 5 years
  Radiation dose (mGy-cm)

CONTACTS AND LOCATIONS:
Overall Officials: Trial Manager, Study Chair — Jinling Hospital, Nanjing University School of Medicine, Nanjing, China.

IPD SHARING:
Plan to Share IPD: No